CLINICAL TRIAL: NCT02263534
Title: Randomized Controlled Trial Comparing Minisling to Tension Free Vaginal Tape in Mangement of Stress Urinary Incontinence
Brief Title: Comparing Minisling to Tension Free Vaginal Tape in Mangement of Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Reda, specialist obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIMS001
Record Dates: First submitted 2014-08-20; First posted 2014-10-13 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; tension free vaginal tape; single incision minisling; midurethral sling
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- minisling (Experimental): patients in this arm will undergo single incision minisling
  Interventions: Procedure: single incision minisling
- tension free vaginal tape (Sham Comparator): patients in this arm will undergo tension free vaginal tape
  Interventions: Procedure: tension free vaginal tape

INTERVENTIONS:
Procedure: single incision minisling — midline incision of the vagina at midurethral level dissection of the vagina from perivesical fascia insertion of the tape (polypropylene macropore mesh tape) in the retropubic direction with its end grasped with an artery forceps till level of perineal membrane closure of the vagina 2 sham incisions if the skin only will be made at suprapubic to maintain blindness posterior colpoperneorraphy will be carried out if needed
  Arms: minisling
Procedure: tension free vaginal tape — midline incision of the vagina at midurethral level dissection of the vagina from perivesical fascia insertion of the tape (polypropylene macropore mesh tape) with the applicators in the retropubic direction and 2 skin incision will be made supra pubic through which the applicators will be passed and removed and the tape will be cut at level just below the skin closure of the vagina posterior colpoperneorraphy will be carried out if needed
  Other Names: TVT
  Arms: tension free vaginal tape

SUMMARY:
Based on previous studies the single incision minisling is an easy less invasive procedure with fewer complications and cure rate similar to conventional midurethral slings in the treatment of female stress urinary incontinence. The aim of this study is to test the hypothesis that the single incision mini-sling placed in the "U" position is not inferior to TVT in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urodynamic stress urinary incontinence, with or without pelvic organ prolapse

Exclusion Criteria:

* Patients with overactive bladder on urodynamic study.
* Patients with voiding dysfunction.
* Patients with intrinsic sphincteric deficiency.
* Patients with previous anti-incontinence surgery.
* Patients on anti-coagulant therapy.
* Immune-compromised patients (DM, patients on corticosteroids treatment).
* Refusal of surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
objective cure rate of urinary incontinence at 12 months after surgery | 12 months
  Objective cure is indicated by a negative stress test and the absence of any additional surgical or nonsurgical treatment for stress urinary incontinence
subjective cure rate of urinary incontinence at 12 months after surgery | 12 months
  subjective cure is indicated by an Incontinence Severity Index score of 0 and the absence of any additional surgical or nonsurgical treatment for stress urinary incontinence

SECONDARY OUTCOMES:
Number of participants with short- term complications | 12 months
  short-term complications (less than 6 weeks): post-operative pain, urinary retention, denovo urgency and wound sepsis
Number of participants with long-term complications | 12 months
  long-term complications: erosion, dyspareunia and recurrence

CONTACTS AND LOCATIONS:
Overall Officials: ahmed reda, M.Sc, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839